CLINICAL TRIAL: NCT06719180
Title: A Prospective Randomized Controlled Trial of Vaginal Cuff Anesthesia and Post-Operative Pain Medication Use
Brief Title: Vaginal Cuff Anesthesia and Post-Operative Pain Medication Use
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: MediSys Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2172359
Record Dates: First submitted 2024-11-22; First posted 2024-12-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hysterectomy; Post Operative Analgesia
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vaginal Cuff Anesthesia (Experimental)
  Interventions: Drug: Bupivacain
- Vaginal Cuff Saline (Placebo Comparator)
  Interventions: Other: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Bupivacain — Injection into the vaginal cuff will occur before vaginal cuff closure with stratafix suture. There will be four points of injection 1cm from the edges of the vaginal cuff with a sterilized needle to a depth of 3-4cm. 5cc of bupivacaine with epinephrine or 5cc of normal saline will be injected into each area
  Arms: Vaginal Cuff Anesthesia
Other: Saline (NaCl 0,9 %) (placebo) — A saline placebo
  Arms: Vaginal Cuff Saline

SUMMARY:
The purpose of this study is to determine whether an injection of a local anesthetic (Bupivacaine with epinephrine) in the vaginal cuff prior to closure would result in less immediate postoperative pain medication and increase patient comfort/satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older requiring total laparoscopic hysterectomy with or without bilateral salpingo-oophorectomy for benign conditions
* Presence of malignancy

Exclusion Criteria:

* Conversion to laparotomy

  * Previous multiple abdominal and/or pelvic surgeries
  * Significant medical comorbidities or cardiac history
  * Poor initial Aldrete score4 (<10)
  * Significant pre-op pain medication use
  * Contraindication to any medication that would be used in the study (Bupivacaine, epinephrine, tramadol or oxycodone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Milligrams of Morphine Equivalent Used | From enrollment to end of treatment at 4 hours.

SECONDARY OUTCOMES:
Counts of Non-Opioid Analgesics Used | From enrollment to end of treatment at 4 hours.
Patient Change in Pain Score (0-10) | From Baseline to end of treatment at 4 hours
  Change in value of pain score, measured on a 0-10 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Flushing Hospital Medical Center, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided